CLINICAL TRIAL: NCT03434873
Title: Effect of Motor Cortex Magnetic Stimulation Versus Sacral Magnetic Stimulation in Lower Urinary Tract Dysfunction in Multiple Sclerosis Patients
Brief Title: Effect of Motor Cortex Versus Sacral Magnetic Stimulation in Multiple Sclerosis Patients With Urinary Tract Dysfunction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, May Maged Abdel-Salhin, Doctor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 30091981
Record Dates: First submitted 2018-02-02; First posted 2018-02-15 (Actual); Last update posted 2018-02-15 (Actual); Status verified 2018-02

CONDITIONS: Multiple Sclerosis; Lower Urinary Tract Symptoms
Keywords: magnetic stimulation, multiple sclerosis
MeSH Terms: conditions — Multiple Sclerosis; Lower Urinary Tract Symptoms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sacral magnetic stimulation (Active Comparator): Twenty trains of 50 stimuli at 5 Hz (train duration: 10 seconds) separated by a 40-second pause were delivered for a total of 1000 pulses, once a day for four consecutive days for two weeks, over sacral roots
  Interventions: Other: magnetic stimulation
- Cortical magnetic stimulation (Active Comparator): Twenty trains of 50 stimuli at 5 Hz (train duration: 10 seconds) separated by a 40-second pause were delivered for a total of 1000 pulses, once a day for four consecutive days for two weeks, over motor cortex
  Interventions: Other: magnetic stimulation

INTERVENTIONS:
Other: magnetic stimulation — Twenty trains of 50 stimuli at 5 Hz (train duration: 10 seconds) separated by a 40-second pause were delivered for a total of 1000 pulses, once a day for four consecutive days for two weeks

SUMMARY:
This work is intended to assess the effect of repetitive magnetic stimulation on the sacral roots versus repetitive magnetic stimulation on motor cortex in multiple sclerosis patients with the lower urinary tract dysfunction.

DETAILED DESCRIPTION:
Twenty Multiple sclerosis patients with lower urinary tract symptoms will be receiving repetitive magnetic stimulation on sacral roots. Another twenty Multiple sclerosis patient with lower urinary tract symptoms will be receiving repetitive magnetic stimulation on motor cortex. Treatment outcome will be assessed and compared between the two groups.

Twenty trains of 50 stimuli at 5 Hz (train duration: 10 seconds) separated by a 40-second pause were delivered for a total of 1000 pulses (total duration: 16 minutes) once a day for four consecutive days for two weeks.

ELIGIBILITY:
Inclusion Criteria:

* Multiple Sclerosis patients (diagnosed by McDonald criteria 2010) with lower urinary tract dysfunction
* Adults more than 18 years
* Unresponsiveness to medical treatment
* Urodynamic diagnosis of detrusor overactivity and/or detrusor underactivity and/or detrusor-sphincter dyssynergia

Exclusion Criteria:

* Urinary tract infections
* Pregnancy

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2014-10; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Change from baseline King's Health QoL questionnaire score after treatment | 1-7 days after treatment
  questionnaire evaluates the impact of lower urinary tract symptoms on patient's quality of life.
  High scores represent a worse quality of life, with no cut-off values.
Change from baseline Post-void residual urine after treatment | 1-7 days after treatment
  Measured by ultrasound It is the volume of urine left in the bladder at the completion of micturition Measured in milliliters (mL)
Change from baseline Maximum Cystometric Capacity (MCC) after treatment | 1-7 days after treatment
  Measured by urodynamic evaluation Measured in millimeters (mL) It is the volume at which the patient states that he/she can no longer delay micturition because of strong desire to void or urgency
Change from baseline Maximum Flow Rate (Qmax) after treatment | 1-7 days after treatment
  Measured by urodynamic evaluation Measured in milliliters per second (mL/sec) It is the maximum measured value of the flow rate
Change from baseline Detrusor pressure at maximum flow rate (Pdet @Qmax) after treatment | 1-7 days after treatment
  Measured by urodynamic evaluation Measured in centimeter water (cmH2O) It represents the effect of the active and/or passive forces generated by the detrusor muscle